CLINICAL TRIAL: NCT05609942
Title: A Phase 1/2, Open-label, 2-arm Study Evaluating BLU-263 as Monotherapy and in Combination With Azacitidine, in Patients With KIT Altered Hematologic Malignancies
Brief Title: Study of Elenestinib (BLU-263) in Advanced Systemic Mastocytosis (AdvSM) and and Other KIT Altered Hematologic Malignancies
Acronym: AZURE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated - alignment of strategic priorities
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BLU-263-2101; 2022-001535-87 (EudraCT Number)
Record Dates: First submitted 2022-11-02; First posted 2022-11-08 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Advanced Systemic Mastocytosis
Keywords: BLU-263; elenestinib; azacitidine; AdvSM; KIT D816V; Advanced systemic mastocytosis; Mast cell leukemia; MCL; Systemic mastocytosis; SM; SM-AHN; CMML-2; Myelodysplastic/myeloproliferative neoplasms; MDS/MPN; Myeloid neoplasms; ASM
MeSH Terms: conditions — Mastocytosis, Systemic; Leukemia, Mast-Cell; Myelodysplastic-Myeloproliferative Diseases | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monotherapy (Experimental): Participants with AdvSM (ASM, SM-AHN, or MCL) will receive BLU-263 monotherapy.
  Interventions: Drug: BLU-263
- Combination therapy (Experimental): Participants with high risk and very high risk systemic mastocytosis with an associated hematologic neoplasm (SM-AHN) of non-MC lineage will receive BLU-263 in combination with azacitidine.
  Interventions: Drug: BLU-263; Drug: Azacitidine

INTERVENTIONS:
Drug: BLU-263 — BLU-263 Oral Tablets
  Other Names: elenestinib
Drug: Azacitidine — Azacitidine powder for suspension for intravenous infusion / subcutaneous injection
  Arms: Combination therapy

SUMMARY:
The goal of this clinical trial is to evaluate elenestinib (BLU-263) in participants with Advanced Systemic Mastocytosis (AdvSM), SM with an associated hematologic neoplasm (SM-AHN), and other hematologic malignancies. The main questions it aims to answer are:

* Determine Recommended Dose of elenestinib (BLU-263) monotherapy for participants with AdvSM
* Safety and tolerability of elenestinib (BLU-263) monotherapy
* Efficacy of elenestinib (BLU-263) monotherapy in participants with AdvSM
* Determine Recommended Dose of elenestinib (BLU-263) in combination with azacitidine in participants with AdvSM
* Safety and tolerability of elenestinib (BLU-263) in combination with azacitidine
* Efficacy of elenestinib (BLU-263) in combination with azacitidine in participants with AdvSM

The estimated study duration for each participant will be approximately 4 years: 2 years of treatment followed by 2 years of follow-up. Participants may be required to attend monthly visits for the first six months, followed by quarterly visits for the remainder of the study.

DETAILED DESCRIPTION:
Systemic mastocytosis includes five major subtypes: Indolent SM (ISM), SM with an associated hematologic neoplasm (SM-AHN), aggressive SM (ASM), and MC leukemia (MCL). In 2016, the smoldering subtype of SM, a former provisional ISM subvariant, was designated as a distinct variant of SM by the World Health Organization (WHO). Aggressive SM, SM-AHN, and MCL together are referred to as Advanced SM (AdvSM).

ELIGIBILITY:
Key Inclusion Criteria :

* Participant has Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2
* Participant must have a new Bone Marrow (BM) biopsy or may use archival tissue if taken within 56 days prior to C1D1 and participant must be willing to have follow-up BM Biopsies.
* Participants receiving antineoplastic therapy within the preceding 12 weeks must have discontinued therapy due to disease progression, refractory disease, lack of efficacy, or intolerance.
* Participants treated with 1 prior selective KIT inhibitor (such as avapritinib or CGT9486) will be permitted on study after confirmation of KIT D816V mutation and with written approval of the study Sponsor. Participants who discontinued treatment with a prior selective KIT inhibitor due to a severe AE that was thought to be related to prior treatment will not be eligible to participate in the study.

Arm 1 (Monotherapy): Participants must have one of the following AdvSM diagnoses, based on World Health Organization (WHO) diagnostic criteria.

Before enrollment, diagnosis of AdvSM must be confirmed based on Central Pathology Laboratory assessment of BM:

1. Aggressive SM (ASM).
2. SM-AHN that in the opinion of the Investigator is not considered to be a candidate for Hypomethylating agent (HMA) monotherapy. Incidental indolent, low-grade lymphoid AHNs (eg, chronic lymphocytic leukemia) not requiring treatment are eligible.
3. Mast cell leukemia (MCL), including diagnoses with an AHN component, that does not require a C-finding.
4. Upon discussion with the Sponsor, other relapsed or refractory hematologic neoplasms with evidence of aberrant KIT or PDGFR may be considered for enrollment. (eg, participants with chronic myeloid neoplasms, such as subvariants of MDS/MPN that harbor activating KIT exon 17 mutations but do not fulfill the diagnostic criteria of SM-AHN, and participants with myeloid/lymphoid neoplasms with PDGFRa/b fusion genes and mutations conferring resistance to imatinib, such as T674I or D842V).

Key Exclusion Criteria:

* Diagnosis of a Philadelphia chromosome positive malignancy
* Acute myeloid leukemia.
* If the participant is receiving corticosteroids, and the dose has not been stable for ≥7 days.
* Within the 14 days prior to enrollment, participant has received any antineoplastic therapy (including midostaurin, avapritinib and other tyrosine kinase inhibitors [TKIs]) or an investigational agent.
* Participant has received hydroxyurea within 7 days prior to the first dose of elenestinib (BLU-263).
* Participant received prior HMA therapy (e.g., azacitidine, decitabine) for the current diagnosis.
* Participant must not be eligible for allogenic hematopoietic stem cell transplantation.
* Participant received prior radiotherapy within 14 days of screening BM biopsy.
* Participant received any hematopoietic growth factor (except erythropoietin) within 14 days of screening BM biopsy, or requiring growth factors to maintain adequate neutrophil or platelet levels.

Those participants maintained on a chronic dose of erythropoietin, whose hemoglobin is stable, and dose of erythropoietin has not been changed in the prior 28 days are allowed on study.

* Participant received >1 prior selective KIT inhibitor (eg: avapritinib or bezuclastinib).
* Participant have any of the following laboratory abnormalities on last laboratory assessment within 14 days prior to the first dose of initiation of study drug: a. Alanine aminotransferase and aspartate aminotransferase > 3 × ULN; > 5 × ULN if associated with clinically suspected liver infiltration by mastocytosis or another disease for which the patient enrolled into the study b. Total bilirubin > 1.5 × ULN; > 3 × ULN if associated with liver infiltration by the disease being treated or in the presence of Gilbert's Disease. (In the case of Gilbert's disease, a direct bilirubin > 2.0 ULN would be an exclusion) c. Estimated (Cockcroft-Gault formula) or measured creatinine clearance < 40 mL/min d. Absolute neutrophil count < 0.5 × 10^9/L
* Participant has had a major surgical procedure within 14 days of the first dose of study drug.
* History of another primary malignancy that has been diagnosed or required therapy within 1 year prior to the first dose of study drug. The following are exempt from the 1-year limit: completely resected basal cell and squamous cell skin cancer, curatively treated localized prostate cancer, GI stromal tumor, and completely resected carcinoma in situ of any site.
* Mean resting QTcF > 480 msec, a history of prolonged QT syndrome or Torsades de pointes, or a familial history of prolonged QT syndrome.
* Clinically significant, uncontrolled, cardiovascular disease.

Arm 1 (Monotherapy):

* Myelodysplastic Syndrome (MDS) that is very high- or high-risk as defined by the International Prognostic Scoring System for Myelodysplastic Syndromes-Revised (IPSS-R).
* A myeloid AHN with ≥10% BM or peripheral blood blasts.
* Platelet count <50 x 10^9/L (within 4 weeks prior to the first dose of study drug) or receiving platelet transfusions or thrombopoietin receptor agonists (TPO-RA) within the prior 14 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Dose Escalation: Number of Dose-limiting Toxicities (DLTs) (monotherapy only) | 28 Days
  Monotherapy: The Recommended Dose (RD) will be primarily determined by the number of DLTs in the first 28 days of treatment with elenestinib (BLU-263) monotherapy.
Dose Escalation: Number of DLTs (combination therapy only) | 28 Days
  Combination therapy: The RD will be primarily determined by the number of DLTs (during 28 days starting from Day 15 of C1 or Day 15 of C2) with elenestinib (BLU-263) in combination with azacitidine.
Dose Escalation and Expansion: Pure Pathological Response (PPR) Rate for SM in Selective KIT Inhibitor-naïve Participants (monotherapy only) | Up to approximately 4 years
  PPR Rate is defined as complete remission (resolution of palpable splenomegaly/hepatomegaly) (CR) + complete remission with partial recovery of peripheral blood counts (CRh) + partial remission (≥35% reduction in spleen volume) (PR)
Dose Escalation and Expansion: Number of Participants with Adverse Events (AEs) | Up to approximately 4 years
Dose Escalation and Expansion: Number of Participants with Serious Adverse Events (SAEs) | Up to approximately 4 years

SECONDARY OUTCOMES:
Dose Escalation and Expansion: Overall Response Rate (ORR) for AdvSM using modified International Working Group-Myeloproliferative Neoplasms Research and Treatment and European Competence Network on Mastocytosis (IWG-MRT-ECNM) (monotherapy only) | Up to approximately 4 years
  ORR is defined as CR + CRh + PR + Clinical Improvement (CI)
Dose Escalation and Expansion: ORR for SM Using Modified IWG-MRT-ECNM (combination therapy only) | Up to approximately 4 years
Dose Escalation and Dose Expansion: Maximum Plasma Concentration (Cmax) of BLU-263 | Up to approximately 4 years
Dose Escalation and Dose Expansion: Cmax of Azacitidine (combination therapy only) | Up to approximately 4 years
Dose Escalation and Dose Expansion: Time to Maximum Concentration (Tmax) of BLU-263 | Up to approximately 4 years
Dose Escalation and Dose Expansion: Tmax of Azacitidine (combination therapy only) | Up to approximately 4 years
Dose Escalation and Dose Expansion: Area Under the Curve From Time Zero to 24 Hours (AUC(0-24)) of BLU-263 | Up to approximately 4 years
Dose Escalation and Dose Expansion: AUC(0-24) of Azacitidine (combination therapy only) | Up to approximately 4 years
Dose Escalation and Dose Expansion: Apparent Volume of Distribution (Vz/F) of BLU-263 | Up to approximately 4 years
Dose Escalation and Dose Expansion: Vz/F of Azacitidine (combination therapy only) | Up to approximately 4 years
Dose Escalation and Dose Expansion: Terminal Elimination Half-life (t1/2) of BLU-263 | Up to approximately 4 years
Dose Escalation and Dose Expansion: t1/2 of Azacitidine (combination therapy only) | Up to approximately 4 years
Dose Escalation and Dose Expansion: Apparent Oral Clearance (CL/F) of BLU-263 | Up to approximately 4 years
Dose Escalation and Dose Expansion: CL/F of Azacitidine (combination therapy only) | Up to approximately 4 years
Dose Escalation and Dose Expansion: Accumulation Ratio of BLU-263 | Up to approximately 4 years
Dose Escalation and Dose Expansion: Accumulation Ratio of Azacitidine (combination therapy only) | Up to approximately 4 years
Dose Escalation and Expansion: Overall Survival (OS) (monotherapy only) | Up to approximately 4 years
Dose Escalation and Expansion: Time to Response (TtR) (monotherapy only) | Up to approximately 4 years
Dose Escalation and Expansion: Duration of Response (DOR) (monotherapy only) | Up to approximately 4 years
Dose Escalation and Expansion: Progression-Free Survival (PFS) (monotherapy only) | Up to approximately 4 years
Dose Escalation and Expansion: Proportion of Participants Pursuing Stem Cell Transplant (monotherapy only) | Up to approximately 4 years
Dose Escalation and Expansion: PPR Rate for SM (combination therapy only) | Up to approximately 4 years

CONTACTS AND LOCATIONS:
Locations (11):
- United States (4):
  - Stanford Cancer Institute, Palo Alto, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Belgium (2):
  - Antwerp University Hospital, Edegem
  - University Hospital Ghent, Ghent
- CHU Caen - Institut d'Hematologie de Basse Normandie, Caen, France
- University Medical Centre Mannheim, Mannheim, Germany
- Maastricht University Medical Center, Maastricht, Netherlands
- Oslo University Hospital, Oslo, Norway
- Instituto de Estudios de Mastocitosis de Castilla La Mancha (CLMast), Toledo, Spain

IPD SHARING:
Plan to Share IPD: No